CLINICAL TRIAL: NCT01660464
Title: Guided Self-Help for Parents of Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD): A Feasibility and Effectiveness Study
Brief Title: Guided Self-Help for Parents of Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Manfred Doepfner, Leading psychologist at the Department of Child and Adolescent Psychiatry, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADHD-Team-03
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Program evaluation; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADHD-Team (Experimental): Intervention
  Interventions: Behavioral: CBT Based Self-help Workbook + Counseling Telepho

INTERVENTIONS:
Behavioral: CBT Based Self-help Workbook + Counseling Telepho — Over a period of 12 months parents work through 8 self-help booklets and additionally receive 14 counseling telephone calls. The intervention has a cognitive-behavioral foundation. Primary purpose of counseling telephone calls is to clarify contents of the booklets and support parents in managing their homework assignments accompanied with each booklet.
  Other Names: Guided self help; behavioral treatment

SUMMARY:
Cognitive-behavioral based guided self-help for parents of adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD) is investigated in a feasibility and effectiveness study. The treatment is offered under routine-care conditions of the health-care system in Germany. Practicability, treatment participation and effectiveness is documented and tested in a one-group pre-test/post-test design.

DETAILED DESCRIPTION:
Self-directed interventions may overcome many of the barriers associated with accessing face-to-face services, as there is lowered stigma and significantly reduced or eliminated cost, transport, and timing difficulties. Families can complete self-directed programs at home, in their own time and at their own pace. Furthermore self-administered programs are often very cost-effective and their use can ease the financial burden of mental health of the community. These parenting programs can be particularly effective by reaching the populace. Moreover in primary care settings where financial resources, time and expertise might be lacking to provide behavioral interventions, self-directed programs might be a promising tool for disseminating effective parenting interventions more widely.

Bibliotherapy is one form of self-directed therapy. In bibliotherapy a selected book is thought to meet the specific need of the person to be treated and reading is used as the therapeutic technique. In opposition to pure self-help programs, bibliotherapy in terms of guided self-help provides patients (or parents) with written instructions as well as therapeutic contacts at regular intervals. During these contacts, problems and questions can be discussed to give further support. Self-help interventions have already proven to be effective for adults with anxiety or affective disorders as well as for depressive adolescents. However there has only been little research concerning the reduction of children's and adolescent´s behaviour problems through parental self-help programs under minimal contact conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent with a diagnosis of ADHD

Exclusion Criteria:

* Language or reading difficulties of participating parent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Total score of the Symptom Checklist Attention-Deficit/Hyperactivity Disorder (SCL-ADHD, Döpfner, Görtz-Dorten & Lehmkuhl, 2008 | 1 year
  Questionnaire assesses the diagnostic criteria of DSM-IV and ICD-10 for ADHD. Informant is participating parent.

SECONDARY OUTCOMES:
Strengths & Difficulties Questionnaire (SDQ) | 1 year
  Questionnaire assesses comorbid symptoms. Informant is the participating parent.
Quality of Life Questionnaire KINDL (Ravens-Sieberer & Bullinger, 2000) | 1 year
  Questionnaire assesses child´s quality of life. Informant is participating parent.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne, Cologne, North Rhine-Westphalia, Germany